CLINICAL TRIAL: NCT01154556
Title: Non-nucleoside Reverse Transcriptase Inhibitor Failure in a High HIV Caseload Australian Primary Care Practice
Brief Title: RETRIeVE: ReversE TranscRiptase Inhibitor hiV Practice
Status: Completed | Type: Observational
Sponsor: Holdsworth House Medical Practice (Other)
Responsible Party: Principal Investigator, Dr. Mark Bloch, Principal Investigator, Holdsworth House Medical Practice
Other Study IDs: RETRIeVE
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: HIV Positive
Keywords: Antiretroviral therapy experienced; failed NNRTI regime
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- HIV1 positive, NNRTI exposure and failure

SUMMARY:
An observational retrospective study of NNRTI experienced patients who have virologically failed. The study aims to assess resistance profiling and subsequent prescription patterns of patients on NNRTIs

DETAILED DESCRIPTION:
This is a cross-sectional study involving retrospective review of HIV-1 positive patient records who began treatment with a non-nucleoside reverse transcriptase inhibitor (NNRTI) and subsequently failed. Patients who have virologically failed previous NNRTI treatment, or have resistance to 1 drug in the NNRTI class are examined further. Such patients will have attended the clinic every 3-6 months for routine medical care. The data source for variables collected is the patient's electronic medical records. This database is located at Holdsworth House Medical Practice (HHMP), Sydney.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV infection
2. Attended Holdsworth House Medical Practice 1999-2009.
3. Chosen ART regime includes an NNRTI

Exclusion Criteria: N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Demographic information will be collected from patient medical records for all patients that have used previously, or are currently using an NNRTI as part of HIV treatment therapy.
Sampling Method: Probability Sample
Enrollment: 2044 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
resistance profiling and subsequent prescription patterns of patients on NNRTIs | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Holdsworth House Medical Practice, Darlinghurst, New South Wales, Australia